CLINICAL TRIAL: NCT02666040
Title: A Multicenter Prospective Randomized Study Of Comparison Between Semi-Absorbable Prosthesis And Totally Nonabsorbable Prosthesis In Inguinal Hernia Surgery
Brief Title: Study on Ultrapro vs Polypropylene: Early Results From a Multicentric Experience in Surgery for Hernia
Acronym: SUPERMESH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Zeta Research Ltd (Industry)
Responsible Party: Principal Investigator, Michele Tedeschi, Clinical Research Coordinator, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-v035
Record Dates: First submitted 2016-01-14; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- U - ULTRAPRO (Experimental): Inguinal Hernia Surgery with ULTRAPRO® meshes, a new ULTRAPRO® mesh will be implanted in patients in the group (AG). The surgery will be evaluated in terms of procedure, detecting the mode of admission to hospital, the duration of surgery, anesthesia volume and type used, composition of the surgical equipment.
  Interventions: Device: ULTRAPRO® meshes; Procedure: Detecting the mode of admission to hospital; Procedure: Duration of surgery; Procedure: Anesthesia volume and type used
- P - Prolene (Active Comparator): Inguinal Hernia Surgery with "Prolene®" meshes, the conventional mesh in polypropylene "Prolene®" will be implanted in patients in the control group (CG). The surgery will be evaluated in terms of procedure, detecting the mode of admission to hospital, the duration of surgery, anesthesia volume and type used, composition of the surgical equipment.
  Interventions: Device: "Prolene®" meshes; Procedure: Detecting the mode of admission to hospital; Procedure: Duration of surgery; Procedure: Anesthesia volume and type used

INTERVENTIONS:
Device: ULTRAPRO® meshes — The inguinal hernia repair has to be performed with the Lichtenstein technique, with standardized prosthesis fixation and no use of plug.
  Arms: U - ULTRAPRO
Device: "Prolene®" meshes — The inguinal hernia repair has to be performed with the Lichtenstein technique, with standardized prosthesis fixation and no use of plug.
  Arms: P - Prolene
Procedure: Detecting the mode of admission to hospital — Ordinary admission or day surgery
Procedure: Duration of surgery — Time operating room
Procedure: Anesthesia volume and type used — Anesthesias used: infiltration, followed by spinal, general, epidural.

SUMMARY:
With reference to inguinal hernia surgeries with prosthesis, the multicenter study aims to investigate the benefits in terms of incidence of pain and discomfort, improvement in the quality of life for the patient after the use of the newly introduced semi-absorbable prosthesis (ULTRAPRO® meshes) compared with the prosthesis of totally nonabsorbable material (conventional meshes in polypropylene "Prolene®"), and in terms of the costs for the hospital, the National Health System (NHS), and the society of associates for the use of the ULTRAPRO® in inguinal hernia surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Males and females
* Adults over 18
* All primitive inguinal hernia

Exclusion Criteria:

* Emergency surgery
* Impossibility to complete the follow-up
* Patients with acquired immunodeficiency symptoms
* Patients with relapsed inguinal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Chronic pain or discomfort evaluated at 6 months, by Visual Analogic Scale for pain (VAS) | 6 months after the operation
  VAS is a horizontal line, 100 mm in length, anchored by word descriptors (no pain, very severe pain) at each end.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montorsi, Prof., Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan